CLINICAL TRIAL: NCT03813888
Title: Effect of Arshvidya After School Program on Cognitive Processes in Elementary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other); Arsha Vidya Study Centre, Tamilnadu, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NMP/ Arsha/0092
Record Dates: First submitted 2019-01-21; First posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Cognitive Change

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arsha Vidya Group (Experimental): After school, children joined regular sessions in Arsha Vidya study centre to practice, vedic chants, vedanta reading, yoga and group activities within the ashram.
  Interventions: Other: Arsha Vidya chldren's Group
- Usual Activity Group (Other): After school, control group were asked to conitue their usual routine.
  Interventions: Other: Usual Activity group

INTERVENTIONS:
Other: Arsha Vidya chldren's Group — Yoga, Vedic chants, Vedant sessions, Gita sessions and group activities within the Gurukulam (centre)
  Arms: Arsha Vidya Group
Other: Usual Activity group — Usual after school activities at home.
  Arms: Usual Activity Group

SUMMARY:
The impact of Arsha Vidya program on cognitive performance was examined in elementary school children. The study compares the effects of arsha vidya after school routine with usual after school routine in healthy 8-11 year-old Indian children.

The main objective of the study is to investigate the effect on cognitive function, behaviour and emotions.

ELIGIBILITY:
Inclusion Criteria:

* Be 8 - 11 years of age at the start of the intervention
* Healthy Children
* Not start new activity within the intervention period
* Parental conset
* Parents to allow and participate where needed in intervention

Exclusion Criteria:

* Serious chronic illnesses and diseases
* Diagnosed with any psychiatric illness
* Intake of medication that may affect study outcomes
* not able to continue for 12-weeks of participation

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Cognitive function | Change from baseline to 12-week
  Cognitive functions measured by the Cambridge Neuropsychological Test Automated Battery

SECONDARY OUTCOMES:
Behaviour | Change from Baseline to 12-weeks
  Behaviour measured by the Behavior Rating Inventory of Executive Function
Attention | Change from baseline to 12-weeks
  Attention measured by the D2 Test of Attention

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Warwick Research Services; Puneet Sharma, Study Director — Sarvatra International, Dubai; Buddhatmananda Saraswati, Study Chair — Arsha Vidya Study Centre, India
Locations (1):
- NMP Medical Research Institue, Jaipur, Rajasthan, India